CLINICAL TRIAL: NCT02168218
Title: Effects of Milk Proteins on Whole Body Protein Synthesis and Ectopic Lipid Deposition During Sucrose Overfeeding in Healthy Male Subjects
Brief Title: Effects of Milk Proteins on Protein Synthesis in Healthy Male Subjects Fed a Hypercaloric, High Sucrose Diet
Acronym: FruMilk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Luc Tappy, MD, Professor of Physiology, University of Lausanne
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 218/13
Record Dates: First submitted 2014-06-05; First posted 2014-06-20 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Obesity
Keywords: protein synthesis; intrahepatic fat; lean body mass; IGF1; energy metabolism
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- high protein (Experimental): 20% protein diet
  Interventions: Other: 7-day overfeeding
- low protein (Active Comparator): 7.5% protein diet
  Interventions: Other: 7-day overfeeding

INTERVENTIONS:
Other: 7-day overfeeding — 7-day overfeeding with an excess sucrose intake corresponding to 40% total energy requirements

SUMMARY:
This study aims at assessing the hypothesis that dietary protein content is a major factor regulating lean body mass gain and energy expenditure during overfeeding, and thus long term body weight gain

To test this hypothesis, healthy normal weight male and female subjects will before and after a 7-day hypercaloric, high-sucrose diet (+40% excess energy as sucrose) and either a low (5% total energy) or a high (20% total energy) protein intake. Each subject will be studied with both low- and high protein diets according to a randomized, crossover study. On each occasion the following measurements will be done in basal conditions (after 2-day isoenergetic, controled diet) and at the end of the 7-day overfeeding:

* whole-body protein turnover, oxidation and synthesis in fasting conditions and fed conditions (13C-labelled leucine)
* intrahepatic and intramuscular fat concentration (1H-Magnetic Resonance Spectroscopy)
* Energy metabolism in fasted and fed conditions (indirect calorimetry)
* plasma concentration of glucose, non-esterified fatty acids, total triglyceride, very-low density lipoprotein (VLDL)-triglyceride, insulin, glucagon, growth hormone (GH), insulin-like growth factor 1 (IGF1), insulin-like growth factor binding protein (IGFBP) 1,2 and 3 in fasting and fed conditions The effects of high-protein and low-protein sucrose overfeeding on whole body protein synthesis will be compared using two-way ANOVA; relationships between changes in whole body protein synthesis on one hand, and intrahepatic/intramuscular fat concentrations, total energy expenditure, and plasma concentration of metabolic variables on the other hand, will be evaluated by linear regression analysis

ELIGIBILITY:
Inclusion Criteria:

* good apparent health
* low physical activity
* non-smokers

Exclusion Criteria:

* vegans or following any special diet
* consumption of > 3 dl/day sweetened beverages
* changes in body > +/- 3Kg over the past 3 months
* contra-indications to magnetic resonance spectroscopy
* drug or substance abuse
* consumption > 10g/day alcohol
* lactose intolerance

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
whole body protein synthesis | after two days of a run-in, isocaloric low sucrose diet and after 7 days of a hypercaloric, high sucrose diet
  Whole body protein synthesis, protein turnover, and protein oxidation will be calculated using 13C-labelled leucine infusion in both fasted and fed conditions

SECONDARY OUTCOMES:
intrahepatic and intramuscular fat concentration | after two days of a run-in, isocaloric low sucrose diet and after 7 days of a hypercaloric, high sucrose diet
  Intrahepatic and intramuscular fat concentration will be measured by in-vivo 1H-Magnetic Resonance Spectroscopy
Energy expenditure | after two days of a run-in, isocaloric low sucrose diet and after 7 days of a hypercaloric, high sucrose diet
  Energy expenditure will be measured by indirect calorimetry min fasted and fed conditions
Metabolic variables in plasma samples | after two days of a run-in, isocaloric low sucrose diet and after 7 days of a hypercaloric, high sucrose diet
  Plasma glucose, insulin, nonesterified fatty acids, triglycerides, VLDL-triglycerides, insulin, glucagon GH, IGF1, IGFBP1, 2 and 3 will be measured in fasted and fed conditions

CONTACTS AND LOCATIONS:
Overall Officials: Luc Tappy, MD, Principal Investigator — University of Lausanne
Locations (1):
- CHUV-clinical research center, Lausanne, Canton of Vaud, Switzerland